CLINICAL TRIAL: NCT06662903
Title: A Comparative Study Between Cranioplasty Using Titanium Mesh Vs Bone Cement
Brief Title: Cranioplasty Using Titanium Mesh Vs Bone Cement
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Osman Hassan Osman Zafraan (Other)
Responsible Party: Sponsor-Investigator, Osman Hassan Osman Zafraan, Resident doctor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cranioplasty
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Bone Defects; Decompressive Craniectomy and Cranioplasty; Cranioplasty
Keywords: Cranioplasty; Titanium mesh; Bone cement; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Bone Cements

STUDY DESIGN:
Intervention Model Description: Titanium mesh VS Bone cement in Cranioplasty
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Titanium mesh (Active Comparator): this group is operated using titanium mesh
  Interventions: Procedure: Cranioplasty with Titanium mesh
- Bone cement (Active Comparator): this group is operated using bone cement
  Interventions: Procedure: Cranioplasty with bone cement

INTERVENTIONS:
Procedure: Cranioplasty with Titanium mesh — Cranioplasty using titanium mesh
  Arms: Titanium mesh
Procedure: Cranioplasty with bone cement — Cranioplasty using bone cement
  Arms: Bone cement

SUMMARY:
The aim of this study is:

To compare the surgical outcomes between titanium mesh and bone cement in cranioplasty.

To assess the complication rates associated with each material. To evaluate patient satisfaction and aesthetic results post-surgery

DETAILED DESCRIPTION:
Cranioplasty is a common neurosurgical procedure performed to repair skull vault defects.

The skull vault defects may result mostly after traumatic injuries as depressed skull fractures, Tumor removal (infiltrating skull bones), decompressive craniectomies, congenital anomalies or inflammatory lesions.

At present, there is no gold standard material for cranioplasty with the use of autologous bone as well as other synthetic materials as bone cement and titanium mesh.

Bone cement is malleable, lightweight, strong, and heat resistant, but it may cause burn injury during the process of its preparation and is used for relatively small defects.

Titanium mesh good mechanical strength, a low infection rate, and an acceptable cost but may cause metal allergy, tissue erosion, implant exposure, and deformity upon application of external force.

Cranioplasty not only provides Brain protection and cosmetic aspects but also, decrease incidence of epilepsy, relief to psychological drawbacks and increases social performance, restoring the dynamics of CSF.

ELIGIBILITY:
* Inclusion Criteria:

  * Patients requiring cranioplasty for a skull defect due to Decompressive Craniectomy, trauma, tumor resection, or congenital issues.
  * All ages .
  * Both sex.
  * Informed consent obtained from all participants.
  * Patient fit for surgery.
* Exclusion Criteria:

  * Patients with active infection at the surgical site
  * Patient Unfit for surgery.
  * Patient refuse consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction using patient ssatisfaction grade | through study completion, an average 1 years
  Patients satisfaction (cosmetic, psychological, neurologic ) measered by validate questionnaire post-opeartive and follow up using Patient satisfaction grade from Excellent to not satisfied

SECONDARY OUTCOMES:
Infection | through study completion, an average 1 years
  follow up rate of post operative infection
Reoperation | through study completion, an average 1 years
  rate of reoperation after using each material a post-operative follow up
CSF leak | through study completion, an average 1 years
  post-operative complication of CSF leak due to changes in Dynamics of CSF flow
complications | through study completion, an average 1 years
  post-operative as hematoma formation , neurologic defict and fits.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mousa M, Eissa S, Raslan M, Abu ElNaga B, Balaha A. Evaluation of three different methods of cranioplasty; a comparative prospective randomized study. Pan Arab Journal of Neurosurgery. 2021;16
- [Background] Andrabi SM, Sarmast AH, Kirmani AR, Bhat AR. Cranioplasty: Indications, procedures, and outcome - An institutional experience. Surg Neurol Int. 2017 May 26;8:91. doi: 10.4103/sni.sni_45_17. eCollection 2017. PMID 28607825
- [Background] Capitelli-McMahon H, Kahlar N, Rahman S. Titanium Versus Autologous Bone-Based Cranioplasty: A Systematic Review and Meta-Analysis. Cureus. 2023 May 26;15(5):e39516. doi: 10.7759/cureus.39516. eCollection 2023 May. PMID 37366436
- [Background] Aydin S, Kucukyuruk B, Abuzayed B, Aydin S, Sanus GZ. Cranioplasty: Review of materials and techniques. J Neurosci Rural Pract. 2011 Jul;2(2):162-7. doi: 10.4103/0976-3147.83584. PMID 21897681
- [Background] Alkhaibary A, Alharbi A, Alnefaie N, Oqalaa Almubarak A, Aloraidi A, Khairy S. Cranioplasty: A Comprehensive Review of the History, Materials, Surgical Aspects, and Complications. World Neurosurg. 2020 Jul;139:445-452. doi: 10.1016/j.wneu.2020.04.211. Epub 2020 May 6. PMID 32387405